CLINICAL TRIAL: NCT03033966
Title: Evaluation of Cerebral Oxygenation and Hemodynamics in Patients With Cerebral Venous Thrombosis
Status: Completed | Type: Observational
Sponsor: Dhritiman Chakrabarti (Other)
Responsible Party: Sponsor-Investigator, Dhritiman Chakrabarti, Assistant Professor, National Institute of Mental Health and Neuro Sciences, India
Organization: National Institute of Mental Health and Neuro Sciences, India (Other)
Other Study IDs: Item No.6.04, Neurosciences
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Cerebral Venous Thrombosis
Keywords: Cerebral Oximetry; Cerebral Venous Thrombosis; Decompressive Craniectomy
MeSH Terms: conditions — Intracranial Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: NIRS based Cerebral Oximetry — Cerebral Oximetric measurement before and after decompressive craniectomy
  Other Names: Equanox, Nonin Medical, Inc. Plymouth, Minnesota, USA

SUMMARY:
Cerebral hypoperfusion and hypoxia are the major determinants of neurological outcomes following acute brain injury as proved in Traumatic Brain Injury/Sub Arachnoid Haemhorrhage literature. How the brain injury affects cerebral oxygenation in patients with CVT is not currently known. Some of the factors that can affect cerebral oxygenation in patients with CVT are Hemoglobin, PO2, PCO2, Cerebral Perfusion Pressure (or MAP) and change in Intracranial Pressure after Decompressive Craniectomy. This study is designed to study how these factors affect cerebral oxygenation and impact of Decompressive Craniectomy on the cerebral oxygenation.

ELIGIBILITY:
Inclusion Criteria:

-Patients diagnosed with cerebral venous thrombosis, undergoing decompressive craniectomy.

Exclusion Criteria:

* Patients on inotropic support
* Systolic blood pressure < 90 mmHg
* Haemoglobin oxygen saturation <95%
* Refusal of consent
* Age <16 and > 65 years
* Known history of diabetes or hypertension
* Pregnancy
* Any contraindication for application of cerebral oximetry sensors

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Cerebral venous thrombosis for Decompressive craniectomy
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2016-02-10 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Ipsilateral Regional Cerebral Oxygen Saturation | From Recruitment till 48 hours postoperative (end of study)
  Measurement of regional cerebral oxygen saturation over ipsilateral frontal lobe before and after decompressive craniectomy with follow up at postoperative 24 and 48 hours.

SECONDARY OUTCOMES:
Contralateral Regional Cerebral Oxygen Saturation | From Recruitment till 48 hours postoperative (end of study)
  Measurement of regional cerebral oxygen saturation over contralateral frontal lobe before and after decompressive craniectomy with follow up at postoperative 24 and 48 hours.
Systolic Blood Pressure | From Recruitment till 48 hours postoperative (end of study)
  Measurement of systolic blood pressure before and after decompressive craniectomy with follow up at postoperative 24 and 48 hours.
Glasgow coma scale score | From Recruitment till 48 hours postoperative (end of study)
  Measurement of Glasgow coma scale score before and after decompressive craniectomy with follow up at postoperative 24 and 48 hours.
Arterial blood gas measurement | From Recruitment till 48 hours postoperative (end of study)
  Arterial blood gas measurement before and after decompressive craniectomy with follow up at postoperative 24 and 48 hours.
Haemoglobin | From Recruitment till 48 hours postoperative (end of study)
  Haemoglobin measurement before and after decompressive craniectomy with follow up at postoperative 24 and 48 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- NIMHANS, Bengaluru, Karnataka, India

IPD SHARING:
Plan to Share IPD: No
May be shared on individual requests